CLINICAL TRIAL: NCT01843218
Title: Erectile Rating During the Treatment of Rectal Cancers Localized. Exploratory Study
Brief Title: Erectile Rating During the Treatment of Rectal Cancers Localized
Acronym: METEORR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IB2008-07
Record Dates: First submitted 2012-11-06; First posted 2013-04-30 (Estimated); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer Stage I
Keywords: Localized rectal cancer in a male patient
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with localized rectal cancer (Other): Assessment (at night) of erctile dysfunction using R/P recording (RIGISCAN® PLUS / polysomonography)
  Interventions: Other: Evaluation of erectile dysfunction

INTERVENTIONS:
Other: Evaluation of erectile dysfunction — Assessment (at night) of erctile dysfunction using R/P recording (RIGISCAN® PLUS / polysomonography)

SUMMARY:
Sexual dysfunction is a common side effect of medical and surgical treatments for rectal cancer. It can manifest as ejaculation disorders or erectile dysfunction. Due to the modesty of both patients and doctors, these disorders are poorly understood and probably underestimated at present. Aim : Objectively assess the presence of erectile dysfunction induced by medical and surgical treatment of rectal cancer three months after surgery. These objective data will be obtained using the RIGISCAN® PLUS system coupled with polysomnographic recording.

DETAILED DESCRIPTION:
Sexual dysfunction is a common side effect of medical and surgical treatments for rectal cancer. It can manifest as ejaculation disorders or erectile dysfunction. Due to the modesty of both patients and doctors, these disorders are poorly understood and probably underestimated at present. After surgical treatment alone, sexual dysfunction can be observed in 40 to 90% of patients, depending on the studies and the technique used. It is the result of direct vascular and nerve damage caused during surgery. It occurs immediately after surgery. It can sometimes recover over time, up to 18 months after the operation. Pelvic radiotherapy also has side effects on sexual function. The damage is caused by alterations in microvascularization or direct nerve damage.

It develops more gradually, over a period of several weeks or months. After treatment combining radiotherapy and surgery, the risk of sexual dysfunction is significant and can affect up to 90% of patients.

In an attempt to improve these results, surgical techniques have gradually evolved towards complete resection of the mesorectum with nerve preservation. Studies published on this subject show an improvement in functional outcomes, without any deterioration in oncological outcomes. This has now become the standard surgical technique.

In the specific case of the management of neoplastic disease, it is common to observe a reactive anxiety-depression syndrome in patients. This mood disorder affects libido and sexuality. A lack of sexual activity in the postoperative period is therefore not necessarily related to iatrogenic vascular-nerve damage. In order to improve patients' quality of life, it is useful to know how to objectively diagnose post-operative erectile dysfunction. This diagnosis should make it possible to distinguish between disorders related to vascular-nervous damage and those that are part of a post-operative anxiety-depression syndrome.

An accurate diagnosis of sexual dysfunction can lead to specific treatment:

intracavernosal injections of prostaglandins are the standard treatment, but phosphodiesterase 5 inhibitors can also be used. For these reasons, it is necessary to develop a method for evaluating objective erectile dysfunction after resection.

The Rigiscan Plus device is a commercially available measurement tool that has received CE certification.

It can be used to assess several parameters of erection: rigidity, intensity, and duration. This measuring device has been validated for the assessment of erectile dysfunction, and normal values have been established in healthy subjects.

Combining these two tests makes it possible to assess the presence or absence of erections during REM sleep and to objectively diagnose erectile dysfunction:

in the presence of decreased libido, nocturnal erections are preserved, whereas they are impaired following vascular-nervous damage. Recording nocturnal erections is useful for assessing erectile dysfunction after rectal surgery in two ways. Preoperatively, it provides objective confirmation that the patient has spontaneous erections of good quality. Postoperatively, recording allows confirmation that the autonomic nervous system required for erection has been preserved. It is an objective examination that is independent of the patient's libido, which is often impaired by the treatment of a neoplastic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male patient.
2. Age greater than 18 years.
3. Neoplastic rectal stage ≤ T3.
4. Patient sexually active before diagnosis.
5. Laparoscopic surgery.
6. Medico-surgical institute Bergonié.
7. Patient information and consent for participation in the study.

Exclusion Criteria:

1. Patients already treated for erectile dysfunction.
2. Absence of sexual activity before diagnosis.
3. Presence of secondary lesions at diagnosis (M +).
4. Classified T4 tumor preoperatively.
5. Surgery by laparotomy.
6. History of pelvic cancer surgery prostate or bladder.
7. History of pelvic radiotherapy (outside of the current process).
8. History of prostate or bladder neoplasia known.
9. Other neoplastic known.
10. Patient for psychological, social, family or geographical could not be treated or monitored regularly according to the criteria of the study, patient deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: EVRARD Serge, PU-PH, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Localized Rectal Cancer
Started | 12
Completed | 7
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Localized Rectal Cancer
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 7

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Erectile Dysfunction Induced by Medical and Surgical Treatment of Rectal Cancer
Description: Erectile dysfunction is defined by the absence of normal nocturnal erections according to R/P recording (RIGISCAN® PLUS / polysomnography)
Time Frame: 3 months after surgery
Population: Participants with R/P recording (RIGISCAN® PLUS / polysomnography) performed
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Localized Rectal Cancer
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Quality of Nocturnal Erections
Description: Erections are assessed according to R/P recording (RIGISCAN® PLUS / polysomnography).
  Erectile function will be described and categorized into 4 distinct stages:
  * Stage 1: Normal erections. Rigidity measured at the tip of the penis is ≥ 60% for at least 10 minutes.
  * Stage 2: Intermediate erections. Rigidity measured at the tip of the penis is between 40 and 60% for at least 5 minutes.
  * Stage 3: Failing erections. Erectile episodes are noted but their intensity is less than 40% OR their duration is less than 5 minutes.
  * Stage 4: Absence of erections. No erectile episodes are recorded.
Time Frame: 3 years after surgery
Population: Participants with available R/P recording (RIGISCAN® PLUS / polysomnography).
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Localized Rectal Cancer
Number analyzed (Participants) | 6
Participants
  Normal erections | 3
  Intermediate erections | 2
  Failing erections | 1
  Absence of erections | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Other [Not Including Serious] Adverse Events were not monitored/assessed for this prospective observational study
Groups:
- Patients With Localized Rectal Cancer: Assessment (at night) of erectile dysfunction using R/P recording (RIGISCAN® PLUS / polysomonography)
  Evaluation of erectile dysfunction: Assessment (at night) of erectile dysfunction using R/P recording (RIGISCAN® PLUS / polysomonography)
Arm/Group | Patients With Localized Rectal Cancer
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes